CLINICAL TRIAL: NCT06948994
Title: A Clinical Trial on Autologous NK Cells Combined With GD2 Monoclonal Antibody in the Treatment of Children With Newly Diagnosed High-risk or Relapsed/Refractory Neuroblastoma
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Guangzhou Women and Children's Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NK-GD2 neuroblastoma
Record Dates: First submitted 2025-04-22; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Neuroblastoma; GD2 Antibody; Autologous NK Cell
Keywords: neuroblastoma; GD2 antibody; autologous NK cell
MeSH Terms: conditions — Neuroblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention arm (Experimental): using autologous NK cells combined with GD2 monoclonal antibody
  Interventions: Combination Product: autologous NK cell plus GD2 antibody

INTERVENTIONS:
Combination Product: autologous NK cell plus GD2 antibody — Combination of autologous NK cells and GD2 monoclonal antibody

SUMMARY:
This is a prospective, single-arm, open, single-center clinical trial to evaluate the safety and efficacy of autologous NK cells combined with chemotherapy and GD2 monoclonal antibody in the treatment of newly diagnosed high-risk or relapsed/refractory neuroblastoma in children. Fifteen eligible subjects are planned to be included. The objective is to evaluate the safety and efficacy of autologous NK cells combined with GD2 monoclonal antibody in the treatment of children with newly diagnosed high-risk or relapsed/refractory neuroblastoma, which is expected to be safe and effective in improving PFS and DCR in children with refractory/recurrent neuroblastoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age 1-18 years (including 18 years), gender not restricted;
2. Diagnosed with high-risk neuroblastoma and meeting the following conditions: high-risk neuroblastoma has undergone standardized treatment including induction therapy and consolidation therapy according to COG, SIOPEN or the expert consensus CCCG-NB-2021, and has entered the maintenance stage; high-risk neuroblastoma has undergone induction therapy with COG chemotherapy combined with GD2 immunotherapy and has entered the maintenance stage; any recurrence of high-risk neuroblastoma after standardized treatment; or the disease is initially determined to be in a refractory state.
3. If it is relapsed/refractory neuroblastoma, there must be at least one measurable lesion according to RECIST 1.1 criteria;
4. Normal major organ function, that is, meeting the following standards:

(1) Blood routine test: hemoglobin >= 80 g/L; absolute neutrophil count (ANC) >=0.75×10^9/L; platelet count >= 75×10^9/L; (2) Blood biochemistry test: serum albumin >=28 g/L; total bilirubin <= 2×upper limit of normal (ULN); aspartate aminotransferase (AST), alanine aminotransferase (ALT) <= 3×ULN; alkaline phosphatase (ALP) <= 3×ULN; creatinine <= 1.5×ULN; (3) Coagulation function: international normalized ratio (INR) or prothrombin time (PT) <= 1.5×ULN; activated partial thromboplastin time (APTT)<=1.5×ULN; (4) Echocardiogram shows normal diastolic function of the heart, left ventricular ejection fraction (LVEF) >= 50%, and no severe arrhythmia; (5) No severe lung or kidney disease, no active pulmonary infection. Indoor air oxygen saturation >=92%; 5. Expected survival time >= 6 months; 6. After obtaining full informed consent from the patient and guardian, sign the informed consent form.

Exclusion Criteria:

1. Uncontrollable active infections, or expected to receive systemic anti-infection or immunosuppressive therapy during participation in this trial;
2. Any toxic reactions caused by previous anti-tumor treatments have not recovered to grade 1 or below (CTCAE 5.0 version) (hair loss is not restricted);
3. Have a history of organ transplantation or are expected to undergo organ transplantation during the trial period;
4. Highly allergic constitution;
5. HIV infection;
6. The researchers believe that there are other circumstances in which the subjects are not suitable to participate in this study.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
adverse event | during the treatment phase
serious adverse event | during the treatment phase
overall survival | 3 years
event-free survival | 3 years

SECONDARY OUTCOMES:
progression-free survival | 3 years

IPD SHARING:
Plan to Share IPD: No